CLINICAL TRIAL: NCT02493465
Title: Effects of Everolimus in Left Ventricular Hypertrophy After Conversion From Azathioprine: A Pilot Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Urologia e Nefrologia (Other)
Responsible Party: Principal Investigator, MARIO ABBUD FILHO, MD PHD, Instituto de Urologia e Nefrologia
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CRAD001ABR33T
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Left Ventricular Hypertrophy
Keywords: everolimus; left ventricular hypertrophy
MeSH Terms: conditions — Hypertrophy, Left Ventricular | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LVH everolimus (Experimental): Progression of left ventricular hypertrophy in recipients of kidney transplant after conversion of immunossupression from azathioprine to everolimus.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Conversion from azathioprine to everolimus in kidneys transplant recipients with left ventricular hypertrophy.

SUMMARY:
This is a prospective, open label, single-center study, in kidney transplant recipients with stable renal function for 12 and 120 months after transplantation, that are in use use of calcineurin inhibitors, azathioprine, and prednisone. The prevalence of left ventricular hypertrophy will be investigated before and after conversion of azathioprine to everolimus.

This study will evaluate as primary objectives: the prevalence of left ventricular mass hypertrophy in renal transplant recipients with azathioprine therapy. And assess the ability of everolimus to reduce left ventricular mass after conversion from Azathioprine, using sensitive methods such as MRI. And as secondaries objectives: Renal function (measured GFR) at 3 and 6 and 12 months after conversion, number and severity of episodes of acute rejection proven by biopsy, and the proteinuria at 3, 6 and 12 months after conversion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (black and white subjects);
* Kidney transplant recipients of living donor or deceased with creatinine clearance (measured / estimated) > 50 ml /L for at least 12 months, receiving azathioprine with or without calcineurin inhibitor with or without prednisone.

Exclusion Criteria:

* The subject, in the opinion of the investigator, is not able to complete the study protocol;
* Multiple organ transplant recipient;
* Pregnant women
* Breastfeeding and childbearing age without contraceptive method
* Test for Positive immunodeficiency virus (HIV)
* Treatment of acute rejection in the last 3 months
* Glomerulonephritis new relapse
* New or polyomavirus nephropathy
* protein / creatinine ≤ 150 mg / mmol or 24h proteinuria> 500mg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Progression of left ventricular hypertrophy | 12 months
  Progression of left ventricular hypertrophy will be mesure by MIR and echocardiography (systolic and end-diastolic diameter of the left ventricle, interventricular septum thickness in end diastole, thickness of the ventricular posterior wall of the left ventricle in end-diastole, left ventricular mass, percentage of left ventricular ejection fraction.

SECONDARY OUTCOMES:
renal function | 3,6, 12 months
  GFR (creatinina clearance)
proteinuria | 3,6, 12 months
  24h Proteinuria
acute rejection episodies | 12 months
  clinical and biopsy if acute rejection suspected

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Urologia e Nefrologia, São José do Rio Preto, São Paulo, Brazil